CLINICAL TRIAL: NCT00388856
Title: Vitamin C and E Supplementation in Pregnant Women With Low Antioxidant Status
Brief Title: Antioxidant Supplementation in Pregnant Women With Low Antioxidant Status
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Showa University (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Yuditiya Purwosunu, Univ. Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17791137
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2007-03

CONDITIONS: Preeclampsia
Keywords: antioxidant supplementation; preeclampsia; prevention
MeSH Terms: conditions — Pre-Eclampsia | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Vitamin C 1000mg and E 400IU

SUMMARY:
The purpose of this study is to investigate antioxidants supplementation in pregnant women with low antioxidant status at 10-12 weeks gestation age in relation to adverse pregnancy outcome in randomized prospective study.

DETAILED DESCRIPTION:
Preeclampsia still remains a leading cause of feto-maternal mortality and morbidity in developed and developing world. Despite of intensive research, the underlying pathologic mechanisms of this disease remain elusive. It has been agreed that incomplete or absent transformation of spiral arteries by replacing endothelial cells and mural vascular smooth muscle cells has been observed in the placental bed of preeclamptic patients and severe cases of intrauterine growth restriction. Oxidative stress has been proposed as a link between these mechanisms. However, it has been demonstrated by two large studies that antioxidant supplementation does not reduce the risk of preeclampsia. Our initial study has been shown that antioxidant supplementation may be reduce the risk of preeclampsia in pregnant women with low antioxidant status.

Comparison(s): adverse pregnancy outcome between vitamin C and E given and placebo given to pregnant women with low antioxidant status at 10-12 weeks gestation age

ELIGIBILITY:
Inclusion Criteria:

* Agree to consent form, and consent to protocol of research
* Known healthy singleton 6-10 weeks pregnant women

Exclusion Criteria:

* Blood pressure > 135/85
* Proteinuria
* History or current use of anti-hypertensive medication or diuretics
* Use of vitamins C > 150 mg and/or E > 75 IU per day
* Pregestational diabetes
* Known placental abnormalities.
* Current pregnancy is a result of in vitro fertilization
* Regular use of platelet active drugs or non-steroidal anti-inflammatory drugs
* Known fetal abnormalities
* Documented uterine bleeding within a week of screening
* Uterine malformations
* History of medical complications
* Illicit drug or alcohol abuse during current pregnancy
* Intent to deliver elsewhere
* Known psychologic problems.
* Participating in another interventional study

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
preeclampsia cases

SECONDARY OUTCOMES:
adverse pregnancy outcome

CONTACTS AND LOCATIONS:
Overall Officials: Akihiko Sekizawa, MD, PhD, Principal Investigator — Showa University School of Medicine
Locations (1):
- Cipto Mangunkusumo National Hospital, Jakarta, Jakarta Special Capital Region, Indonesia